CLINICAL TRIAL: NCT02027649
Title: K14 in Urothelial Cells as a Pronostic and Diagnostic Marker in Bladder Cancer Patients Using a Non Invasive Technique.
Brief Title: Detection of K14 in Bladder Cancer With a Non Invasive Technique
Status: Terminated | Type: Observational
Why Stopped: Absence of positive results
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Juan Francisco Delgado de la Poza, Medical Doctor, Corporacion Parc Tauli
Other Study IDs: K14 in bladder cancer; CIR2013 (Other Grant/Funding Number: Fundació Parc Taulí)
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Keratin 14; Pronostic marker; Diagnostic marker; Noninvasive technique
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Bladder cancer: Patients who suffered a bladder cancer
- Control group: Patients with urologic diseases of non tumoral origin

SUMMARY:
By an invasive technique keratin 14 has been identified as a prognostic factor in bladder cancer. This study aims to analyze whether through a non-invasive technique keratin 14 can be used as a diagnostic and prognostic marker for this cancer.

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer

Exclusion Criteria:

* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Keratin 14 | At the time of study entry

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitària i Universitària Parc Taulí, Sabadell, Barcelona, Spain